CLINICAL TRIAL: NCT01817192
Title: A Randomized Prospective Trial of Adjuvant Chemotherapy in Patients With Completely Resected Stage I or IIA Non-Squamous Non-Small Cell Lung Cancer Identified as Intermediate or High Risk by a 14-Gene Prognostic Assay
Brief Title: Adjuvant Chemotherapy in Patients With Intermediate or High Risk Stage I or Stage IIA Non-squamous Non-Small Cell Lung Cancer: AIM-HIGH (Adjuvant Intervention in Molecular High Risk Patients)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Razor Genomics (Industry)
Collaborators: Encore Clinical (Other)
Responsible Party: Sponsor
Organization: Encore Clinical (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-120888; IFCT-2002 (Other: The French Cooperative Thoracic Intergroup)
Record Dates: First submitted 2013-03-16; First posted 2013-03-25 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Squamous; Adjuvant Chemotherapy; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Participant
Masking Description: Results of 14-Gene prognostic assay will not be revealed to the patient. Low risk patients will be observed, intermediate and high risk patients will be randomized to observation or four cycles of a platinum-based doublet therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation (Active Comparator): Post-operative observation of Stage I or Stage IIA non squamous non-small cell lunger cancer with Radiographic Surveillance is a current standard of care. Patients identified as low risk will be observation. Those patients identified as intermediate or high-risk by the 14-Gene Prognostic Assay will be randomized either to this arm or the Adjuvant Chemotherapy Arm.
  Interventions: Other: Radiographic surveillance; Other: 14-Gene Prognostic Assay
- Adjuvant Chemotherapy (Active Comparator): Adjuvant Chemotherapy is a current standard of care for intermediate or high-risk Stage I or Stage IIA non-squamous non-small cell lung cancer. Patients identified as intermediate or high-risk by the 14-Gene Prognostic Assay will be randomized either to this arm or the Observation Arm.
  Interventions: Drug: Adjuvant Chemotherapy; Other: 14-Gene Prognostic Assay

INTERVENTIONS:
Drug: Adjuvant Chemotherapy — Patients who have undergone complete resection of NSCLC that has been documented histologically to be non-squamous and that is pathological Stage I or IIA, will undergo testing with the 14-Gene Prognostic Assay. Patients determined to be intermediate or high risk and who meet all eligibility criteria will be randomized either to observation or to four cycles of adjuvant therapy with a standard NSCLC platinum-based doublet.
  Arms: Adjuvant Chemotherapy
Other: Radiographic surveillance — Serial radiographic surveillance is a current standard of care for Stage I or Stage IIA lung cancer. All intermediate or high risk patients randomized to observation or chemotherapy will have routine CT Scans at 6 month intervals until 5 years after enrollment and at yearly intervals thereafter until the end of the study period.
  Arms: Observation
Other: 14-Gene Prognostic Assay — This CLIA-approved assay is a standard tool that is now available to all clinicians to improve the prognostic evaluation of patients after resection of Stage I or Stage IIA non-squamous NSCLC. It will be performed on tumor specimens for patients who are potentially eligible for this study. Patients identified through the assay as intermediate or high-risk will be randomized to either adjuvant chemotherapy or observation.

SUMMARY:
The optimal treatment for Stage I or Stage IIA non-small cell lung cancer (NSCLC) remains controversial. Radiographic surveillance alone has been recommended for stage I and stage IIA patients after the tumor is removed surgically from the lung, and this standard has been based on the fact that no previous clinical trial has demonstrated a benefit for Stage I or Stage IIA NSCLC patients who receive post-operative chemotherapy. These patients, however, have a substantial risk of death within five years after operation, ranging from approximately 30% to 45%, largely due to metastatic disease that is present immediately after surgery but that is undetectable by conventional methods. Some leading organizations therefore currently recommend post-operative chemotherapy as an alternative standard of care in Stage I or Stage IIA NSCLC patients who are considered to be at particularly high-risk. Up until now, however, there has not been a well-validated means to identify stage I and stage IIA NSCLC patients at high risk of death within five years after operation. A new prognostic tool, a 14-Gene Prognostic Assay, which has been validated and definitively demonstrated in large scale studies to identify intermediate and high-risk stage I or Stage IIA patients with non-squamous NSCLC, is now available to all clinicians through a CLIA-certified laboratory. It is therefore now possible to compare the outcomes of patients randomly assigned to one or the other of these competing standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Able to comply with the protocol, including acceptable candidacy for adjuvant chemotherapy according to local institutional standards and likely compliance with follow-up for anticipated length of study (i.e. 5 years from the initiation of enrollment).
* Willing to be randomized to chemotherapy.
* Histologically documented completely resected (R0) Stage I or IIA non-squamous NSCLC (per 8th edition, TNM staging system)
* Adequate tissue sample for the 14-Gene Prognostic Assay
* Life expectancy excluding NSCLC diagnosis ≥ 5 years
* ECOG performance status 0-1

Exclusion Criteria:

* Final pathologic diagnosis of pure squamous cell, pure small cell, or pure neuroendocrine histology, or any combination of only these three histologies
* Evidence of greater than stage IIA pathologic staging
* Evidence of incomplete resection
* Pregnant or lactating women
* Unwilling to use an effective means of contraception
* Active infection, either systemic or at site of primary resection
* Systemic chemotherapy or anti-cancer agent within 5 years prior to enrollment
* Radiotherapy to the chest in the immediate pre- or post- operative period
* Malignancies other than the current NSCLC within 5 years prior to randomization, except for adequately treated CIS of the cervix, non-melanoma skin cancer, localized prostate cancer treated locally, ductal carcinoma in situ treated surgically
* Treatment with any investigational drug or participation in another clinical trial within 28 days prior to enrollment
* Known hypersensitivity to study treatment agents
* Evidence of any other disease including infection that contraindicates the use of systemic cytotoxic chemotherapy or puts the patient at high risk for treatment-related complications
* Wound dehiscence or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | 5 years
  To compare Disease Free Survival in patients with resected, stage I or IIA non-squamous NSCLC found to be at intermediate or high risk by the 14-Gene Prognostic Assay randomized to either observation or adjuvant therapy with 4 cycles of a platinum-based doublet.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  To compare Overall Survival in patients randomized to each study arm. To further document the previously verified separation of the survival curves among high and low risk patients identified by the 14-Gene Prognostic Assay in this prospective cohort of stage I or IIA non-squamous NSCLC.

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Principal Investigator — Sarah Cannon, The Cancer Institute of HCA Healthcare
Locations (49):
- United States (18):
  - Leonard Cancer Institute, Mission Viejo, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Providence Medical Foundation Santa Rosa, Santa Rosa, California
  - Sarah Cannon- FCS South, Fort Meyers, Florida
  - Sarah Cannon- FCS North, Petersburg, Florida
  - Sarah Cannon- FCS Panhandle, Tallahassee, Florida
  - Sarah Cannon- FCS East, West Palm Beach, Florida
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Mercy Hospital Joplin Missouri, Joplin, Missouri
  - Mercy Oncology Research St. Louis, St Louis, Missouri
  - Hackensack Meridian Health, Neptune City, New Jersey
  - Sarah Cannon- Messino Cancer Center, Asheville, North Carolina
  - Mercy Oncology Research Oklahoma City, Oklahoma City, Oklahoma
  - Allegheny Health Network Research Institute, Pittsburgh, Pennsylvania
  - St. Francis Cancer Center, Greenville, South Carolina
  - Sarah Cannon Tennessee Oncology, Nashville, Tennessee
  - Swedish Cancer Institute, Seattle, Washington
- France (23):
  - Polyclinique Bordeaux Nord, Bordeaux, Cedex
  - Hôpital Charles Nicolle, Rouen, Cedex
  - CHU d'Angers Service Pneumologie, Angers
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHRU Besançon- Hôpital J. MINJOZ, Besançon
  - Hôpital APHP Ambroise Paré, Boulogne
  - Hia Percy, Clamart
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital Europeen, Marseille
  - Hôpital Nord, Marseille
  - Groupe Hospitalier Région de Mulhouse Sud -Alsace, Mulhouse
  - Centre Hospitalier Universitaire de Nîmes, Nîmes
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Hôpital Paris Saint Joseph, Paris
  - Hôpital Bichat, Paris
  - Hôpital Haut-Lévèque (Bordeaux - CHU), Pessac
  - Chu de Poitiers, Poitiers
  - Hôpital Larrey, Toulouse
  - CHRU de Tours, Tours
  - Gustave Roussy, Villejuif
- Germany (8):
  - Köln-Merheim, Cologne
  - München-Gauting, Gauting
  - Niels-Stensen-Kliniken, Georgsmarienhütte
  - Lung Clinic Grosshansdorf-Department of Thoracic Oncology, Großhansdorf
  - Medizinische Hochschule Hannover, Hanover
  - University Medical Center Schleswig-Holstein, Lübeck
  - University Hospital of Munich, München
  - Pius-Hospital Oldenburg Medizinischer Campus Universität Oldenburg, Oldenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kratz JR, He J, Van Den Eeden SK, Zhu ZH, Gao W, Pham PT, Mulvihill MS, Ziaei F, Zhang H, Su B, Zhi X, Quesenberry CP, Habel LA, Deng Q, Wang Z, Zhou J, Li H, Huang MC, Yeh CC, Segal MR, Ray MR, Jones KD, Raz DJ, Xu Z, Jahan TM, Berryman D, He B, Mann MJ, Jablons DM. A practical molecular assay to predict survival in resected non-squamous, non-small-cell lung cancer: development and international validation studies. Lancet. 2012 Mar 3;379(9818):823-32. doi: 10.1016/S0140-6736(11)61941-7. Epub 2012 Jan 27. PMID 22285053
- [Background] Woodard GA, Wang SX, Kratz JR, Zoon-Besselink CT, Chiang CY, Gubens MA, Jahan TM, Blakely CM, Jones KD, Mann MJ, Jablons DM. Adjuvant Chemotherapy Guided by Molecular Profiling and Improved Outcomes in Early Stage, Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2018 Jan;19(1):58-64. doi: 10.1016/j.cllc.2017.05.015. Epub 2017 May 31. PMID 28645632
- [Background] Kratz JR, Van den Eeden SK, He J, Jablons DM, Mann MJ. A prognostic assay to identify patients at high risk of mortality despite small, node-negative lung tumors. JAMA. 2012 Oct 24;308(16):1629-31. doi: 10.1001/jama.2012.13551. No abstract available. PMID 23093159
- [Derived] Spigel DR, Westeel V, Anderson IC, Greillier L, Guisier F, Bylicki O, Badin FB, Rousseau-Bussac G, Deldycke C, Griesinger F, Bograd A, Zhong W, Le Treut J, Van Hulst S, Gandara DR, Reck M, Hoffknecht P, Gubens MA, Crowley J, von der Leyen H, Woodard GA, Jablons DM, Kratz JR, Mann MJ; AIM-HIGH investigators. Adjuvant chemotherapy for stage IA-IIA non-squamous, non-small-cell lung cancer identified as molecular high-risk by a 14-gene expression profile (AIM-HIGH): an international, randomised, phase 3 trial. Lancet Respir Med. 2025 Oct;13(10):887-896. doi: 10.1016/S2213-2600(25)00213-9. Epub 2025 Jun 24. PMID 40578381